CLINICAL TRIAL: NCT01033058
Title: Effect of Intensive Statin Treatment on 90-day Prognosis of STEMI Patients Undergoing Emergency Primary PCI Compared With Usual Care
Brief Title: Intensive Statin Treatment for STEMI Patients Undergoing Primary PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Prof. Yang Xinchun, Beijing Chaoyang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN2009CV005
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-11

CONDITIONS: STEMI
Keywords: STEMI; atorvastatin; PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (Active Comparator)
  Interventions: Drug: atorvastatin
- intensive statin treatment (Experimental)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — 80mg atorvastatin immediately after enrollment, emergency PCI,atorvastatin 40mg/d and other usual medication after PCI
  Other Names: Lipitor
  Arms: intensive statin treatment
Drug: atorvastatin — No loading dose of statin after enrollment, emergency PCI, atorvastatin 20mg/d and other usual medication after PCI
  Other Names: Lipitor
  Arms: usual care

SUMMARY:
This is a retrospective, randomized, parallel, open-labeled, controlled study to find out whether STEMI patients undergoing emergency PCI can benefit from intensive atorvastatin treatment compared with routine treatment.

DETAILED DESCRIPTION:
ARMYDA-ACS, ARMYDA-RECAPTURE and NAPLES II demonstrated that in patients with ASP and NSTE ACS undergoing early PCI, loading dose of atorvastatin before early PCI led to a reduction of prei-PCI MI, recurrent CV events and mortality. While, theses studies included patients with non-ST-segment elevation ACS, requiring PCI; these results cannot be extrapolated directly to patients with ST-segment elevation MI, and these trials included patients sent to an early and selective PCI, but not those undergoing emergency revascularization;

This study is designed to find out whether STEMI patients undergoing emergency PCI can benefit from intensive atorvastatin treatment compared with routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years old
* myocardiac ischemia symptom of index event appeared less than 12 hours before enrollment.
* ECG showed elevated ST segment in 3 or more contiguous leads
* diagnosed with acute STEMI
* eligible for primary PCI, and primary PCI is scheduled within 2 hours after enrollment

Exclusion Criteria:

* allergic or experienced serious adverse reaction to HMG-CoA reductase
* pregnancy, lactation, or child bearing potential women without any effective contraception
* accompanied with malignant disease
* active hepatic disease or hepatic dysfunction

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The combined endpoint of 90-day all cause morality, cardiac death, recurrent MI, recurrent symptomatic myocardiac ischemia, target vessel revascularization | 2009 Dec- 2011 Mar

CONTACTS AND LOCATIONS:
Overall Officials: Xinchun Yang, Prof., Principal Investigator — Beijing Chaoyang Hospital, China
Locations (1):
- Chaoyang Hospital, Beijing, Chaoyang, China